CLINICAL TRIAL: NCT05950542
Title: Evaluation of Safety and Efficacy of Topical Baricitinib Plus Excimer Light Versus Excimer Light Alone in Treatment in Non-Segmental Vitiligo
Brief Title: Evaluation Safety ,Efficacy Baricitinib Plus Excimer Light Versus Excimer Light Alone in Non Segmental Vitiligo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noura Mohamed Aboud Tawfik, General practitioner physician, Assiut University
Other Study IDs: Baricitinib versus Excimer
Record Dates: First submitted 2023-07-07; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Vitiligo, Generalized
MeSH Terms: conditions — Vitiligo | interventions — baricitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Vitiligo lesions on the face will be treated with cream (Olumiant)2mg twice daily and excimer light308nm DEKA, Florence,Italy twice weekly for 12 weeks.
  Interventions: Drug: Baricitinib
- Group B: Vitiligo lesions on the face will be treated with excimer light308nm (DEKA,F lorence,Italy) only twice weekly for 12 weeks.

INTERVENTIONS:
Drug: Baricitinib — JAK inhibit0rs
  Other Names: Excimer light308nm
  Groups: Group A

SUMMARY:
The study aims to evaluate the safety and efficacy of the combination of topical baricitinib and 308-nm monochromatic excimer light versus 308-nm monochromatic excimer light alone in treatment of non-segmental vitiligo.

DETAILED DESCRIPTION:
Vitiligo is an acquired pigmentary skin disorder characterized by the absence of pigmentary cells from the epidermis that results in white macules and patches on the body. (1) The pathogenesis of vitiligo is unknown, but an autoim¬mune hypothesis prevails. (2, 3) CD8+ inflammatory damage induced by cytotoxic T cells is one of the key immune responses leading to depigmentation and destruction of melanocytes in vitiligo. (4-6) The IFN-γ - chemokine (CXCL9/10-CXCR3) axis, with its associated positive feedback loop, has been identified as a potential pathway in the initiation and progression of the immune response in vitiligo via inhibiting melanogenesis, inducing apoptosis of melanocytes, and further recruiting CD8+ T cells to the skin. (7-9) Janus kinases (JAKs) are a family of cytoplasmic tyrosine kinases (TYKs). (10) They aid cytokine-mediated signal transduction through the JAK/STAT pathway. (11) The key members of this unique tyrosine kinase family include JAK1, JAK2, JAK3, and TYK2. (12) The IFN-γ signaling is dependent on the JAK/STAT pathway. IFN-γ activates the JAK/STAT1 pathway, especially through JAK1 and JAK2. (13) This leads to the phosphorylation of STAT1, with subsequent transcription of IFNγ-induced genes, namely CXCL9 and CXCL10. (14) Given the role of JAK1 and JAK2 in the JAK/STAT pathway, IFN-γ signals can be blocked by inhibiting JAK1 or JAK2. (15) The treatment of vitiligo is generally and challenging, moreover, the goal of treatment is not only to halt disease progression, but promote repigmentation. (16) There are a variety of therapeutic possibilities including topical, systemic and surgical methods encompass grafting and transplantation. (17) The 308 nm excimer laser represents the latest alternative NB-UVB therapy for treating vitiligo. It's a gas laser that can emit a wavelength of 308 nm UVB produced by xenon and chlorine gases. (18) The effectiveness and safety of 308 nm excimer laser phototherapy are superior to that of NB-UVB phototherapy, which may be explained by the ability of the excimer laser to emit coherent pulses, as well as differences in phototherapeutic parameters, such as impulse frequency and intensity, therapy stimulating a deeper reservoir of melanocytes in hair follicles. (19) JAK inhibitors can block the IFN-γ signaling via the JAK-STAT pathway and thus have become an emerging treatment for vitiligo. (20) Based on clinical trials, the US Food and Drug Administration (FDA) approved topical Ruxolitinib 1.5%, a JAK 1 and 2 inhibitor, in patients 12 years of age or older for the treatment of non-segmental vitiligo. (21) In the treatment of vitiligo, a few published case reports, case series, and open-label studies have shown superior re-pigmentation rates in patients treated with JAK inhibitors, especially with concomitant ultraviolet or sun exposure. (22) Given IFN-γ signaling is specially mediated by JAK1 and JAK2, baricitinib, a newer JAK1 and JAK2 inhibitor, has been supposed to be effective in treating vitiligo. (23) The effectiveness of oral baricitinib in treating vitiligo has been reported in small case studies. (23-25) Some clinical studies have confirmed that the application of JAK inhibitors can have side effects, such as infection, malignancy, and major adverse cardiovascular events (MACEs). (26) Clinical disease screening of patients before the use of JAK inhibitors and continuous monitoring during their use are essential. (27) Topical administration of the drug results in improved drug delivery, fast onset of action, and the targeted distribution of the active medication to skin lesions while minimizing the safety concerns related to oral administration. Therefore, some experts believe that topical application show better effects and lower adverse reactions. (28, 29) Given the reported effectiveness of oral barcitinib in vitiligo as well as the successful results of topical forms of other JAK inhibitors, we expect that baricitinib would have similar effect if used topically.

ELIGIBILITY:
Inclusion Criteria:

Patients of age above 12y old. Patients with active non-segmental vitiligo, having minimum of 1% body surface area (BSA) affected, with significant facial involvement (≥0.5% of the BSA on the face).

Co-operative patients, agree to join the study and will give consent.

Exclusion Criteria:

Patients receiving phototherapy or any form of systemic therapy for vitiligo during the previous 2 months preceding the study.

Patients applying topical medications to the face during the last month before the study Pregnant or lactating females. Patients with history of allergy to JAK inhibitors, or history of photosensitivity or post inflammatory hyperpigmentation.

Patients with active skin infection at site of treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: cooperation, agreement to join the study , Above 12 years old ,active non segmental vitiligo patients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
F VASI score | 6 months
  Face Vitiligo Aera Scoring Index (F-VASI) score will be calculated at baseline, every 4 weeks during the first 12 weeks (duration of treatment) and 3 months after stopping treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin mostafa Tawfik, Doctor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Phan K, Phan S, Shumack S, Gupta M. Repigmentation in vitiligo using janus kinase (JAK) inhibitors with phototherapy: systematic review and Meta-analysis. J Dermatolog Treat. 2022 Feb;33(1):173-177. doi: 10.1080/09546634.2020.1735615. Epub 2020 Apr 2. PMID 32096671